CLINICAL TRIAL: NCT03574597
Title: SELECT - Semaglutide Effects on Cardiovascular Outcomes in People With Overweight or Obesity
Brief Title: Semaglutide Effects on Heart Disease and Stroke in Patients With Overweight or Obesity
Acronym: SELECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX9536-4388; 2017-003380-35 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1200-5564 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Participants will receive semaglutide as an adjunct to standard-of-care. Estimated trial duration for an individual subject is from 31 to 59 months.
  Interventions: Drug: Semaglutide
- Placebo (semaglutide) (Placebo Comparator): Participants will receive placebo (semaglutide) as an adjunct to standard-of-care. Estimated trial duration for an individual subject is from 31 to 59 months.
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Semaglutide will be injected into a skin fold, in the stomach, thigh or upper arm once a week at the same day of the week (to the extent possible) throughout the trial. Subjects will start semaglutide treatment at 0.24 mg; dose will gradually be increased every 4 weeks up to 2.4 mg.
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Placebo will be injected into a skin fold, in the stomach, thigh or upper arm once a week at the same day of the week (to the extent possible) throughout the trial. Participants will receive placebo at an equivalent dose to semaglutide.
  Arms: Placebo (semaglutide)

SUMMARY:
The researchers are doing the study to see if semaglutide may reduce the risk of having cardiovascular events in patients with overweight or obesity and with prior cardiovascular disease. The participant will either get semaglutide (active medicine) or placebo ("dummy" medicine). Which treatment the participants get is decided by chance. The participant's chance of getting semaglutide or placebo is the same. The participant will get the study medicine in a pen. The participants will need to use the pen to inject the study medicine in a skinfold once a week. The study will last for about 2.5 to 5 years. Participants will have up to 25 clinic visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age greater than or equal to 45 years at the time of signing informed consent
* Body mass index (BMI) greater than or equal to 27 kg/m^2
* Have established cardiovascular (CV) disease as evidenced by at least one of the following: prior myocardial infarction; prior stroke (ischemic or haemorrhagic stroke); or symptomatic peripheral arterial disease (PAD), as evidenced by intermittent claudication with ankle-brachial index (ABI) less than 0.85 (at rest), or peripheral arterial revascularization procedure, or amputation due to atherosclerotic disease

Exclusion Criteria:

Cardiovascular-related:

* Any of the following: myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within the past 60 days prior to the day of screening
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Presently classified as being in New York Heart Association (NYHA) Class IV heart failure

Glycaemia-related:

* HbA1c greater than or equal to 48 mmol/mol (6.5 %) as measured by the central laboratory at screening
* History of type 1 or type 2 diabetes (history of gestational diabetes is allowed)
* Treatment with glucose-lowering agents within 90 days before screening
* Treatment with any glucagon-like-peptide-1 receptor agonist (GLP-1 RA) within 90 days before screening

General safety:

* History or presence of chronic pancreatitis
* Presence of acute pancreatitis within the past 180 days prior to the day of screening
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma
* End stage renal disease or chronic or intermittent haemodialysis or peritoneal dialysis
* Presence or history of malignant neoplasms within the past 5 years prior to the day of screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed
* Severe psychiatric disorder which in the investigator's opinion could compromise compliance with the protocol
* Known or suspected hypersensitivity to trial products or related products
* Previous participation in this trial. Participation is defined as randomisation
* Receipt of any investigational medicinal product within 30 days before screening
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method
* Any disorder, unwillingness or inability, which in the investigator's opinion, might jeopardise the participant's safety or compliance with the protocol

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17604 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept.2834), Study Director — Novo Nordisk A/S
Locations (833):
- United States (205):
  - Central Alabama Research, Birmingham, Alabama
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Healthscan Clinical Trials,LLC., Montgomery, Alabama
  - Synexus Clinical Research US, Inc./Tatum, Glendale, Arizona
  - Synexus Clinical Research, Glendale, Arizona
  - Synexus Rsch /Cnt Phnx Med C, Phoenix, Arizona
  - National Heart Institute Cal, Beverly Hills, California
  - FDRC, Costa Mesa, California
  - Valley Clinical Trials, Covina, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - First Valley Medical Group, Lancaster, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Long Beach VA healthcare System, Long Beach, California
  - Angel City Research, Inc., Los Angeles, California
  - VAGLAHS Clinical Research Center (CRC), Los Angeles, California
  - Riverside University Health System Medical Center, Moreno Valley, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Western University of Health Sciences, Pomona, California
  - Quartz Hill Walk-in Medical Group, inc., Quartz Hill, California
  - TriWest Research Associates, San Diego, California
  - San Diego Family Care, San Diego, California
  - Mills-Peninsula Medical Center, San Mateo, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Encompass Clinical Research_Spring Valley, Spring Valley, California
  - Lundquist Inst-Biomed Innovtn, Torrance, California
  - Synexus Clinical Research US, Inc._Horsham, Vista, California
  - University of Colorado Hospital, Aurora, Colorado
  - Optumcare Colorado Springs, LLC, Colorado Springs, Colorado
  - Optumcare Colorado Springs, Colorado Springs, Colorado
  - New West Physicians,Inc., Golden, Colorado
  - Optumcare Colorado Springs, LLC_Monument, Monument, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Excel Med Ctr Clinical Trials, Boca Raton, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Nature Coast Clin Rsrch_Crystal River, Crystal River, Florida
  - Florida Premier Cardiology, Delray Beach, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Integrative Research Assoc Inc, Fort Lauderdale, Florida
  - Clinical Research of Hollywood_Hollywood, Hollywood, Florida
  - Est Cst Inst for Rsrch,Jksnvil, Jacksonville, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Baptist Heart Specialists_Jacksonville, Jacksonville, Florida
  - Baptist Heart Specialists_Jacksonville Beach, Jacksonville Beach, Florida
  - Reyes Clinical Research, Inc, Miami, Florida
  - International Research Associates, LLC_Miami, Miami, Florida
  - AdventHealth Diab Inst, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - East Coast Institute for Research LLC, Saint Augustine, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Cardio Partners Clin Res Inst, Wellington, Florida
  - Ellipsis Group, Alpharetta, Georgia
  - NSC Research, Inc, Johns Creek, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Family Health Care Center, Statesboro, Georgia
  - Herman Clinical Research LLC, Suwanee, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Apex Medical Research Inc, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Macoupin Research Group, Gillespie, Illinois
  - Chicago Medical Research LLC, Hazel Crest, Illinois
  - Lemah Creek Clinical Research, Oakbrook Terrace, Illinois
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - NorthShore Univ Hlth Sys, Skokie, Illinois
  - Central Illinois Diabetes and Clinical Research, Springfield, Illinois
  - Community Clinical Research_Anderson, Anderson, Indiana
  - American Health Network of Indiana, LLC_Avon_0, Avon, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - American Health Network of IN LLC_Franklin, Franklin, Indiana
  - American Health Network of Indiana, LLC_Greenfield, Greenfield, Indiana
  - Franciscan Health Michigan City, Michigan City, Indiana
  - American Health Network of IN LLC, Muncie, Indiana
  - American Health Network of Indiana, LLC, New Albany, Indiana
  - Velocity Clinical_Valparaiso, Valparaiso, Indiana
  - University of Iowa Prev Inter Ctr, Iowa City, Iowa
  - The University Of Kansas Medical Center - Cray Dia, Kansas City, Kansas
  - Midwest Heart & Vasc Spec, Overland Park, Kansas
  - Cotton O'Neil Clin Research Ctr, Topeka, Kansas
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Norton Clinical Research Group, Louisville, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Louisiana Heart Center, Hammond, Louisiana
  - Barnum Medical Research, Inc., Natchitoches, Louisiana
  - Louisiana Heart Center_Slidell, Slidell, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University Of Maryland School of Medicine, Baltimore, Maryland
  - Ascension Saint Agnes Heart Ca, Baltimore, Maryland
  - MedStar Good Samaritan Hosp, Baltimore, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Centennial Medical Group, Elkridge, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Endo And Metab Cons, Rockville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - ClinSite LLC., Canton, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Belzoni Clinical Research, Belzoni, Mississippi
  - Amicis Centers of Clinical Research, St Louis, Missouri
  - St Louis Heart & Vascular, P.C., St Louis, Missouri
  - Mercury Street Medical Group, PLLC_Butte, Butte, Montana
  - VA NEB - Western IA Health Stm, Omaha, Nebraska
  - University of NE Med Ctr, Omaha, Nebraska
  - Synexus Clinical Research US, Henderson, Nevada
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Southern NH Diabetes and Endo_Nashua, Nashua, New Hampshire
  - UniMed Center, East Brunswick, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Albany Medical College - Endo, Albany, New York
  - Dr. Alexander Perkelvald, Brooklyn, New York
  - Long Island Cardiovascular Consultants PC, Lake Success, New York
  - NYU Grossman School of Med, New York, New York
  - NYU School of Medicine, New York, New York
  - Comprehensive Weight Ctrl Prog, New York, New York
  - Saratoga Clinical Research, Saratoga Springs, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Great Lakes Medical Research, Westfield, New York
  - UNC Eastowne Clinical Trials Unit, Chapel Hill, North Carolina
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Duke University_Durham, Durham, North Carolina
  - Durham VA Medical Center - Duke University, Durham, North Carolina
  - WakeMed Garner Hlthplx, Garner, North Carolina
  - Physician's East Endocrinology, Greenville, North Carolina
  - Duke University - S.E Cardio, Lumberton, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Accellacare, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - The Carl & Edyth Lindner Center, Cincinnati, Ohio
  - Cleveland Clinic_Cleveland, Cleveland, Ohio
  - Providence Health Partners Ctr, Dayton, Ohio
  - Advanced Med Res Maumee, Maumee, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - Corvallis Clinic PC Clinical Research Department, Corvallis, Oregon
  - Oregon Health & Science Uni, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Doylestown Hospital Pharmacy, Doylestown, Pennsylvania
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Richard M Kastelic MD Assoc, Johnstown, Pennsylvania
  - Hospital of the Univ PA, Philadelphia, Pennsylvania
  - Tristar Clin Investigations, PC, Philadelphia, Pennsylvania
  - Parkside Family Medicine, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians Inc., Pittsburgh, Pennsylvania
  - Internal Medicine Associates of Anderson, Anderson, South Carolina
  - Synexus Clin Res US-Anderson, Anderson, South Carolina
  - Medical Uni of SC Charleston, Charleston, South Carolina
  - Palmetto Clinical Research, Greenville, South Carolina
  - Accellacare US Inc._SC, Mt. Pleasant, South Carolina
  - Holston Medical Group Pc, Bristol, Tennessee
  - The Stern Cardiovascular Group, Germantown, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - InvestiClin Research, Nashville, Tennessee
  - MidState Endocrine Associates, Nashville, Tennessee
  - Trinity Clinical Research LLC, Tullahoma, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Arlington Family Res. Ctr Inc, Arlington, Texas
  - Texas Diab & Endo, P.A., Austin, Texas
  - UT Health University of Texas, Bellaire, Texas
  - Thyroid, Endocrinology, and Diabetes, PA, Dallas, Texas
  - Texas Health Physicians Group_Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Northwest Houston Cardiology, P.A., Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Research Institute Of Dallas, Plano, Texas
  - Quality Research Inc, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - San Antonio Prem Int Med, San Antonio, Texas
  - Physician PrimeCare Research Institute, PLLC dba, San Antonio, Texas
  - Audie L. Murphy Va Hospital, Stvhcs, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Houston Center for Clinical Research LLC, Sugar Land, Texas
  - Christus Heart and Vascular Institute, Tyler, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Wade Family Medicine, Bountiful, Utah
  - Kalo Clinical Research, West Valley City, Utah
  - U. of Vermont Med Ctr Burlington, South Burlington, Vermont
  - Inova Cardiology - Mt. Vernon, Alexandria, Virginia
  - Cardiology Consultants of Danville Inc., Danville, Virginia
  - Inova Cardiology-Fairfax, Fairfax, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Strelitz Diabetes Of Eastern V., Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - National Clin Res Inc., Richmond, Virginia
  - VA Medical Center_Salem, Salem, Virginia
  - Bayview Physician Services, Virginia Beach, Virginia
  - Sentara Medical Group_Norfolk, Virginia Beach, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Amherst Family Practice P.C., Winchester, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
  - Confluence Health Hospital, Wenatchee, Washington
  - St. Vincent Hosp-Prevea Health, Green Bay, Wisconsin
  - Clinical Inv Spec, Inc.Kenosha, Kenosha, Wisconsin
  - Aspirus Research Institute, Wausau, Wisconsin
- Algeria (5):
  - Cardiology department CHU Mustapha Pacha. Algiers, Algiers
  - Centre National De la Médecine du Sport, Algiers
  - CHU Issad Hassani, Beni Messous, Cardiology department, Algiers
  - CHU - Hussein dey Cardiology department Nafissa Hamoud, Algiers
  - Cardiology department, Benaouda Benzerdjeb CHU Oran, Oran
- Argentina (10):
  - Instituto de Cardiología de Corrientes, Corrientes, Buenos Aires
  - Fundacion Favaloro, CABA, Buenos Aires, Argentina
  - Sanatorio Güemes, CABA, City of Buenos Aires
  - Centro de Investigación y Prevención Cardiovascular, CABA
  - Centro Médico MEDEOS, CABA
  - Glenny Corp. S.A, CABA
  - Clínica Adventista Belgrano, CABA
  - Medical Center of Diabetes and Nutrition, CABA
  - Instituto Médico DAMIC, Córdoba
  - Sanatorio Plaza, Rosario
- Australia (13):
  - The Canberra Hospital_Garran, Garran, Australian Capital Territory
  - Gosford Hospital, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
  - Advara HeartCare, Milton, Queensland
  - Core Research Centre, Milton, Queensland
  - Cholesterol Care Australia, Wollongabba, Queensland
  - Royal Adelaide Hospital Cardiovascular Clinical Trials, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Monash Cardiovascular Research Centre, Clayton, Victoria
  - Geelong Cardiology Research Unit, Geelong, Victoria
  - Austin Health, Metabolic Disorders Centre, Heidelberg Heights, Victoria
  - HeartCare WA (Joondalup), Joondalup, Western Australia
- Austria (7):
  - Universitätsklinik für Innere Medizin, Graz
  - Univ.-Klinik für Innere Medizin I, Innsbruck
  - LKH Salzburg Universitätsklinikum, Salzburg
  - Klinik Landstraße, Vienna
  - Ordination Dr. Hanusch, Vienna
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Hietzing, Vienna
- Belgium (7):
  - Algemeen Stedelijk Ziekenhuis - Aalst - Interventional Cardiology, Aalst
  - Imeldaziekenhuis - Bonheiden - Department of Endocrinology, Bonheiden
  - CUB Hôpital Erasme_Brussels_1, Brussels
  - Ziekenhuis Oost-Limburg AV - Cardiology, Genk
  - UZ Gent - Cardiology, Ghent
  - UZ Gent_Gent_4, Ghent
  - Jessa Ziekenhuis - Hasselt - Cardiology, Hasselt
- Brazil (15):
  - Cárdio Pulmonar da Bahia, Salvador, Estado de Bahia
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Eurolatino Medical Research Center, Uberlândia, Minas Gerais
  - Cline Research Center, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica S/S, Curitiba, Paraná
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - AngioCor Blumenau, Blumenau, Santa Catarina
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - CIP Centro Integrado de Pesquisas do Hospital de Base, São José do Rio Preto, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Departamento de Gastroenterologia - HCFMUSP, São Paulo, São Paulo
  - Instituto do Coração - HCFMUSP, São Paulo, São Paulo
  - Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
- Bulgaria (16):
  - Medical Centre Diamedical-2013, Dimitrovgrad
  - MHAT Lukovit, Department of Internal Diseases, Lukovit
  - "MHAT - Pazardzhik" AD, Second Department of Internal Diseas, Pazardzhik
  - "UMBAL-Dr. Georgi Stranski" EAD, First Clinic of cardiology, Pleven
  - "UMHAT "Sveti Georgi" EAD, Plovdiv
  - Medical centre Razgrad OOD, Razgrad
  - "MHAT "NCH" EAD, Cardiology clinic, Noninvasive diag. dep., Sofia
  - "MHAT "NCH" EAD, Clinic of Cardiology, Depart. of Cardiology, Sofia
  - "Acibadem City Clinic MHAT Tokuda" EAD,Cardiology department, Sofia
  - "Acibadem City Clinic UMHAT" EOOD, Sofia, Cardiology clinic, Sofia
  - "Diagnostic - Consulting Center Aleksandrovska" EOOD, Sofia
  - "UMHAT "Aleksandrovska" EAD, Cardiology clinic, Sofia
  - "UMHAT "Tsaritsa Yoanna-ISUL"" EAD, Clinic of Cardiology, Sofia
  - "UMHATEM N.I. Pirogov" EAD, Sofia
  - "UMHAT "Sveta Anna" Sofia" AD, Clinic of Cardiology, Sofia
  - "Diagnostic - Consulting Center "Ekvita"" EOOD, Varna
- Canada (28):
  - University of Calgary, Calgary, Alberta
  - C-endo Diab Endo Clin Calgery, Calgary, Alberta
  - Synergy Wellness Clinic, Sherwood Park, Alberta
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Manna Research Inc. (Burlington N), Burlington, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - St. Joseph's Health Care, London, Ontario
  - Manna Research Ottawa, Nepean, Ontario
  - North York Diagn & Cardiac Ctr, North York, Ontario
  - Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Medical Associates of Port Perry, Port Perry, Ontario
  - HHI Research Inc., Scarborough Village, Ontario
  - Manna Research Stoney Creek, Stoney Creek, Ontario
  - The Port Arthur Clinic Research Program, Thunder Bay, Ontario
  - Manna Research Inc._Toronto, Toronto, Ontario
  - ViaCar Recherche Clinique Inc, Brossard, Quebec
  - Manna Research Quebec, Lévis, Quebec
  - Manna Research Mirabel, Mirabel, Quebec
  - Clinique Sante Cardio MC, Montreal, Quebec
  - IRCM, Montreal, Quebec
  - Applied Med Inf Res, Montreal, Quebec
  - Centricity Res Pointe-Claire, Pointe-Claire, Quebec
  - Clin des Mal Lipid de Quebec, Québec, Quebec
  - Ctr Méd. et pro d l'Ost d port, Saint-Marc-des-Carrieres, Quebec
  - Centre de recherché du CHUS, Sherbrooke, Quebec
  - Centre de santé et de services, Terrebonne, Quebec
  - Institut universitaire de cardiologie, Québec
- Colombia (7):
  - Rodrigo Botero S.A.S, Medellín, Antioquia
  - IPS Centro Cientifico Asistencial Jose Luis Accini SAS, Barranquilla, Atlántico
  - Unidad de Estudios Clínicos de la Fundación Cardiovascular de Colombia, Bucaramanga-piedecuesta, Valle Del Menzuli - Santander, Santander Department
  - Fundacion del Caribe para la Investigacion Biomedica-BIOS, Barranquilla
  - Clinica de la Costa, Barranquilla
  - Centro de Investigacion Clinica Avanzada y Multidisciplinari, Medellín
  - CardiovidCentro Cardiovascular Colombiano ClinicaSantaMaria, Medellín
- Croatia (7):
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - Specijalna bolnica Krapinske Toplice - Kardiologija, Krapinske Toplice, Krapinsko Zagorska County
  - Klinicki bolnicki centar Osijek, Osijek
  - KBC Rijeka, Zavod za kardiomiopatije, Rijeka
  - KBC "Sestre milosrdnice", Kardiologija, Zagreb
  - KBC Zagreb, Klinika za bolesti srca i krvnih zila, Zagreb
  - Klinicka bolnica Sveti Duh, Zagreb
- Czechia (12):
  - Fakultni poliklinika, Prague, Czech Republic
  - Edumed Broumov, Broumov
  - Ordinace pro choroby srdce, Chomutov
  - Fakultni nemocnice Hradec Kralove_Hradec Kralove_0, Hradec Králové
  - Nemocnice Jihlava Kardiologie, Jihlava
  - Kardiologické centrum, Liberec
  - Policska nemocnice, Polička
  - Endocare, Prague
  - ResTrial, Prague
  - Nemocnice Slany Kardiologie, Slaný
  - Svitavska nemocnice Kardiologie, Svitavy
  - Vseobecna kardiologicka ambulance, Tábor
- Denmark (6):
  - Herlev og Gentofte Hospital, Hellerup, Capital Region
  - Aalborg Universitetshospital Kardiologisk Afdeling, Aalborg
  - Aarhus Universitetshospital, Skejby Hjertesygdomme, Aarhus N
  - Regionshospitalet Gødstrup, Hjertesygdomme, Herning
  - Hvidovre Hospital Hjertemedicinsk, Hvidovre
  - Kardiologisk Odense & Svendborg, Svendborg
- Finland (7):
  - StudyCor, Jyväskylä
  - Health Step Finland Oy, Kuopio
  - Päijät-Häme Central Hospital, Lahti
  - OYS Sisätautien tutkimusyksikkö, Oulu
  - Seinäjoen keskussairaala, Seinäjoki
  - TAYS Sydänsairaala, Tampere
  - TYKS Sydänkeskus, Turku
- France (17):
  - CHRU Besançon, Besançon
  - Hôpital Jean Verdier, Bondy
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Universitaire de Dijon-Hopital Le Bocage, Dijon
  - Chu Du Bocage, Dijon
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon-1, La Tronche
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Centre Hospitalier de Narbonne, Narbonne
  - CHU de Nice, Nice
  - Aphp-Hopital La Pitie Salpetriere-2, Paris
  - Ap-Hp-Hopital Europeen Georges Pompidou, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Ap-Hp-Hopital Bichat-Claude Bernard-2, Paris
  - Centre Hospitalier Universitaire de Bordeaux-Hopital Haut Leveque-2, Pessac
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-1, Saint-Herblain
  - Les Hopitaux Universitaires de Strasbourg-Hopital Civil-2, Strasbourg
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (31):
  - Universitaetsklinikum Aachen AöR, Aachen
  - Kardiologische Praxis, Bad Homburg
  - Klinische Forschung Berlin (kfgn), Berlin
  - Emovis GmbH, Berlin
  - Synexus Berlin, Berlin
  - Synexus Bochum, Bochum
  - Klinische Forschung Dresden, Dresden
  - Hausaerztlich-Kardiologisches MVZ Am Felsenkeller GmbH, Dresden
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung GmbH, Essen
  - Synexus Frankfurt, Frankfurt
  - MVZ CCB Frankfurt Und Main-Taunus GbR, Frankfurt
  - Denger, Friedrichsthal, Friedrichsthal
  - Klinische Forschung Hamburg, Hamburg
  - Wendisch/Dahl Hamburg, Hamburg
  - Klinische Forschung Hannover, Hanover
  - Chevts, Karlsruhe
  - Appel, Kassel
  - Universitätsklinikum Leipzig, Endokrinologie und Nephrologie, Leipzig
  - AmBeNet GmbH, Leipzig
  - Die Praxis am Ludwigsplatz, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Dr. Axthelm Christoph, Pirna, Pirna
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
  - Steindorf, Schkeuditz, Schkeuditz
  - Klinische Forschung Schwerin, Schwerin
  - Jacob, Villingen-Schwenningen, Villingen-Schwenningen
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
  - Al-Zoebi, Wermsdorf
  - Forschungszentrum Ruhr KliFoCenter GmbH, Dr. med. Kahrmann, Witten
- Greece (14):
  - University Hospital of Athens ATTIKON, Haidari-Athens, Attica
  - Onassis Cardiac Surgery Center, Athens
  - "Laiko" General Hospital of Athens, Athens
  - Hippokration Hospital, Athens
  - Alexandra General Hospital, Therapeutic Clinic, Athens
  - Konstantopouleio G.H. of Athens, "Agia Olga", Athens
  - "Hygeia" General Hospital of Athens, Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - General Hospital of Chios "Skilitsio", Chios
  - University General Hospital of Ioannina,Internal Medicine, Ioannina
  - General Hospital of Lamia, Lamia
  - Univ Gen Hospital Larisa, Cardiology Medicine Clinic, Larissa
  - AHEPA General University Hospital, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
- Hungary (6):
  - Lausmed Kft., Baja, Bács-Kiskun county
  - Szegedi Tudomanyegyetem St Györgyi Albert Klinikai Központ, Szeged, Csongrád-Csanád
  - Léda Platán Magánklinika, Zalaegerszeg, Zala County
  - Debreceni Egyetem Klinikai Központ Belgyógyászati Klinika, Debrecen
  - Bugát Pál Kórház, Gyöngyös
  - Markusovszky Egyetemi Oktatókórház, Szombathely
- India (34):
  - Ramesh Hospitals, Vijayawada, Andhra Pradesh
  - Apex Heart Institute, Ahmedabad, Gujarat
  - CIMS- Care Institute of Medical Sciences, Ahmedabad, Gujarat
  - Shri B. D. Mehta Mahavir Heart Institute, Surat, Gujarat
  - Unicare heart institute and research centre, Surat, Gujarat
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Medanta - The Medicity Multi-Speciality Hospital, Gurugram, Gurgaon, Haryana
  - Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bangalore, Karnataka
  - St John's Medical College Hospital, Bengaluru, Karnataka
  - Kamalnayan Bajaj Hospital, Aurangabad, Maharashtra
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Lokmanya Tilak Municipal Medical College & General Hospital, Mumbai, Maharashtra
  - Holy Family Hospital and Medical Research Centre, Mumbai, Maharashtra
  - Arneja Heart & Multispeciality Hospital, Nagpur, Maharashtra
  - Shri Krishna Hrudayalaya & Critical Care Centre, Nagpur, Maharashtra
  - Vijan Hospital & Research Centre, Nashik, Maharashtra
  - Grant Medical Foundation, Pune, Maharashtra
  - Batra Hospital and Medical Research Center, New Delhi, National Capital Territory of Delhi
  - Maulana Azad Medical College, Delhi, New Delhi
  - All India Institute of Medical Sciences, New Dehli, New Delhi
  - VMMC & Safdarjung Hospital, New Dehli, New Delhi
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - SP Medical College, Bikaner, Rajasthan
  - The Madras Medical Mission, Chennai, Tamil Nadu
  - G Kuppuswamy Naidu Memorial Hospital, Coimbatore, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Vellore, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - Guru Nanak CARE Hospitals, Hyderabad, Telangana
  - Gandhi Memorial Hospital- King George's Medical University, Lucknow, Uttar Pradesh
  - B M Birla Heart Research Centre, Kolkata, West Bengal
  - Narayana Hrudayalya Institute of Cardiac Sciences, Bangalore
  - St John's Medical College and Hospital, Bangalore
  - Dr. BL Kapur Memorial Hospital, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
- Ireland (6):
  - Mater Miscericordiae Hospital, Dublin, Leinster
  - Connolly Hospital, Dublin, Leinster
  - The Heartbeat Trust, Dublin
  - St Vincent's Private Hospital, Dublin
  - Tallaght Hospital - Cardiology, Dublin
  - Mallow Primary Healthcare Centre, Mallow
- Israel (12):
  - Outpatient Diabetes Clinic Soroka MC, Beersheba
  - Diabetes and obesity center of excellence, Rambam MC, Haifa
  - Diabetes Unit Hadassah Ein Karem MC, Jerusalem
  - Hadassah Ein Kerem MC - Cardio, Jerusalem
  - Clinical Research Unit Meir Medical Center, Kfar Saba
  - Institute of Diabetes, Western Galilee MC Nahariya, Nahariya
  - Rabin Medical Center - Hasharon Hospital, Dept. D, Petah Tikva
  - Kaplan MC, Rehovot
  - Cardio Vascular Research Center Sourasky MC, Tel Aviv
  - Institute of Endocrinology, metabolism and hypertension, Tel Aviv
  - Endrocrinolgy Clinic - Sheba Medical Center, Tel Litwinsky
  - Sheba Medica Center - Clinical Research Unit, Tel Litwinsky
- Italy (24):
  - Ospedale Santa Maria Goretti - UOD Diabetologia, Latina, LT
  - Centro di Alta Spec. Diet., Educ. Alim. e Prev. Cardio Metab, San Donato Milanese (MI), MI
  - Pol. Uni. Campus Biomedico UOC Endocrinologia e Diabetologia, Roma, RM
  - AO Papa Giovanni XXIII USS Dietologia Clinica, Bergamo
  - A. O. Universitaria S.ORSOLA-MALPIGHI - U. O. Endocrinologia, Bologna
  - ARNAS Ospedale Garibaldi, Catania
  - Università degli studi G. D'Annunzio Chieti Pescara - CAST, Chieti Scalo
  - Ospedale di San Fermo della Battaglia, Como
  - Azienda Osp-Univ Ferrara-Dip Scienze Mediche-Endocrinologia, Cona - Ferrara
  - AOU Careggi Dipartimento Medico Geriatrico SOD Diabetologia, Florence
  - U.O.D. Dietetica e Nutrizione Clinica, Genova
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
  - Azienda Ospedaliera di Padova Clin.Med.3, Padua
  - Unità Funzionale di nutrizione clinica cod 58.01.3, Palermo
  - IRCCS Fondazione "S. Maugeri" U.O. Medicina Interna ed Endo, Pavia
  - Azienda Ospedaliero Universitaria Pisana Ospedale Cisanello, Pisa
  - UOC di Medicina Interna - Centro Medico dell'Obesità, Roma
  - Policlinico Universitario AGemelli DH Patologie dell'Obesità, Rome
  - Ist.Clinico Humanitas Endocrinologia e Malattie del ricambio, Rozzano (MI)
  - Centro di Alta Spec. Diet., Educ. Alim. e Prev. Cardio Metab, San Donato Milanese (MI)
  - Osp. Santissima Annunziata ASL CN1 Endocrinol. Diabetol., Savigliano (CN)
  - IRCCS Multimedica, Sesto San Giovanni (MI)
  - A.O.U. Senese Policlinico "Le Scotte" , U.O.C. Diabetologia, Siena
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
- Japan (49):
  - Seiwa Clinic, Adachi-ku, Tokyo
  - Toyooka Chuo Hospital, Asahikawa, Hokkaido
  - The Univ. of Tokyo Hp., Dept. of Cardiovascular Medicine, Bunkyo-ku, Tokyo
  - New Tokyo Heart Clinic_Matsudo-shi, Chiba,, Chiba
  - Fukuokaken Saiseikai Futsukaichi Hospital_Cardiovascular Medicine, Chikushino-shi, Fukuoka
  - Ehime Prefectural Central Hospital, Ehime
  - Chiba Tokushukai Hospital, Funabashi-shi, Chiba
  - Gifu Heart Center, Gifu-city, Gifu
  - Hirakata Kohsai Hospital, Hirakata-shi, Osaka
  - Medical Corporation JR Hiroshima Hospital, Hiroshima-shi, Hiroshima
  - Hiroshi Yamaguchi Clinic, Kagoshima-shi, Kagoshima
  - H.E.C Science Clinic, Kanagawa
  - Kasugai Municipal Hospital, Kasugai-shi, Aichi
  - Sugiura Clinic, Kawaguchi-shi, Saitama
  - Steel Memorial Yawata Hospital, Kitakyushu-shi, Fukuoka
  - Chikamori Hospital, Kochi-shi, Kochi
  - Saiseikai Kumamoto Hospital, Kumamoto-shi, Kumamoto
  - Uji Tokushukai Medical Center, Kyoto
  - Koseikai Takeda Hospital, Kyoto-shi, Kyoto
  - Ijinkai Takeda General Hospital, Cardiovascular Medicine, Kyoto-shi,Kyoto
  - Ijinkai Takeda General Hospital, Neurosurgery, Kyoto-shi,Kyoto
  - Medical Corporation Matsuyama-heartcenter Yotsuba Circulatio, Matsuyama-shi, Ehime
  - Shinden Higashi Clinic_Miyagi, Miyagi
  - Shiga General Hospital, Moriyama-shi, Shiga
  - Nagoya Ekisaikai Hospital, Nagoya-shi, Aichi
  - Naha City Hospital, Naha-shi, Okinawa
  - Takagi hospital, Internal Medicine, Okawa-shi, Fukuoka
  - Okayama Medical Center, Okayama-shi, Okayama
  - Takatsuki Red Cross Hospital, Osaka
  - Sakurabashi Watanabe Advanced Healthcare Hospital, Osaka-city, Osaka
  - Saga University Hospital, Department of Cardiology, Saga-shi, Saga
  - Shinsapporo Seiryou Hospital, Intenal Medicine, Sapporo-shi, Hokkaido
  - Hanaoka Seishu Memorial Hospital, Sapporo-shi, Hokkaido
  - Medical corporation Sanseikai Miyanomori Memorial Hospital, Sapporo-shi, Hokkaido
  - Sendai Kousei Hospital_Sendai-shi, Miyagi, Sendai-shi, Miyagi
  - National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - Japan Community Health care Organization Ritsurin Hospital, Takamatsu-shi, Kagawa
  - Kagawa Prefectural Central Hospital, Cardiovascular Medicine, Takamatsu-shi, Kagawa
  - Kagawa Prefectural Central Hospital, Takamatsu-shi, Kagawa
  - Kan-etsu chu-oh Hospital, Takasaki-shi, Gunma
  - Tokorozawa Heart Center, Tokorozawa-shi, Saitama
  - Saino Clinic, Tokorozawa-shi,Saitama
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Fukuwa Clinic, Tokyo
  - Tokyo Shinagawa Hospital Social Medical Corporation Association Tokyokyojuno-kai, Tokyo
  - Minamino Cardiovascular Hospital, Tokyo
  - National Hospital Organization Saitama National Hospital, Wako-city, Saitama
  - Nagata Hospital, Yanagawa-shi, Fukuoka
  - Yokosuka General Hospital Uwamachi, Cardiology, Yokosuka-shi, Kanagawa
- Latvia (8):
  - Ari Med, Daugavpils
  - Meissana Ltd, Liepāja
  - Teterovska practice, Ogre
  - Stradini Cardiology, Riga
  - Medical Centre Pulss 5, Riga
  - Adoria, Riga
  - Health Centre-4, Riga
  - Ziemelkurzeme Regional Hospital, Ventspils
- Malaysia (13):
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Seri Manjung, Seri Manjung, Perak
  - Sarawak Heart Centre, Kota Samarahan, Sarawak
  - University Technology MARA (UiTM) - Puncak Alam, Sungai Buloh, Selangor
  - Klinik Kesihatan Masjid Tanah, Alor Gajah
  - Hospital Sultanah Bahiyah, Alor Star
  - Sarawak Heart Centre, Kota Samarahan
  - National Heart Institute, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Putrajaya, Putrajaya
  - Hospital Queen Elizabeth II, Sabak Bernam
- Mexico (9):
  - CIMAB SA de CV, Torreón, Coahuila
  - Centro de Investigacion Clinica Endocrinologica de Jalisco, Guadalajara, Jalisco
  - Instituto Nacional de Cardiología Ignacio Chavez, Mexico City, México, D.F.
  - Hospital Universitario Dr. José Eleuterio González_Monterrey, Monterrey, Nuevo León
  - Unidad Biomedica Avanzada Monterrey, Monterrey, Nuevo León
  - Centro de atención e investigación cardiovascular del Potosí, San Luis Potosí City, San Luis Potosí
  - Centro para el Desarrollo de la Medicina y la Asistencia, Culiacán, Sinaloa
  - Centro de Investigación Cardiometabólica de Aguascalientes, Aguascalientes
  - Lahoja Asociación para la Investigación y Farmacovigilancia, Durango
- Netherlands (10):
  - Gelre Ziekenhuizen Apeldoorn, Apeldoorn
  - Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - UMC Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Alrijne Leiderdorp, Leiderdorp
  - Bravis Ziekenhuis, Roosendaal
  - Franciscus Gasthuis en Vlietland, Rotterdam
  - D & A Research B.V., Sneek
  - Ziekenhuis Rivierenland Tiel, Tiel
- Norway (9):
  - Ålesund Sjukehus - Hjertemedisinsk poliklinikk, Ålesund
  - Haukeland Universitetssykehus, Bergen
  - Falck Norge AS, Hamar
  - Sykehuset Innlandet Lillehammer, Lillehammer
  - Akershus Universitetssykehus, Nordbyhagen
  - Rikshospitalet - Kardiologisk forskning, Oslo
  - Oslo universitetssykehus HF Ullevål, Oslo
  - Oslo universitetssykehus Aker, Oslo
  - Senter for sykelig overvekt i Helse Sør-Øst, Tønsberg
- Poland (22):
  - NZOZ "CenterMed Lublin" Sp. z o.o., Lublin, Lublin Voivodeship
  - ETG Siedlce, Siedlce, Masovian Voivodeship
  - ETG Warszawa, Warsaw, Masovian Voivodeship
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych, Bialystok, Podlaskie Voivodeship
  - Kresmed Sp. z o. o., Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - PRATIA Centrum Medyczne, Gdynia, Pomeranian Voivodeship
  - Centrum Zdrowia Metabolicznego, Poznan, Wielkopolskie Voivodeship
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - Centrum Badan Klinicznych PI-House, Gdansk
  - Grazyna Pulka Specjalistyczny Osrodek "All-Med", Krakow
  - UniCardia & UniMedica & UniEstetica, Krakow
  - Centrum Terapii Wspolczesnej, Lodz
  - ETG Lowicz, Lowicz
  - Centrum Medyczne HCP Sp. z o.o., Poznan
  - Velocity Nova Sp. z o.o., Puławy
  - Gabinety Lekarskie LabMed, Szczecin
  - Przychodnia Lekarzy Specjalistow Serce, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
  - Velocity Zamość, Zamość
  - Klimed Lomza, Łomża
  - Clinmedica Research sp. z o.o., Skierniewice, Łódź Voivodeship
- Portugal (6):
  - Hospital Garcia de Orta, Almada
  - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Unidade Local de Saúde de Matosinhos, Matosinhos Municipality
  - Centro Hospitalar de São João, Porto
- San Miguel Medical, Trujillo Alto, Puerto Rico
- Romania (26):
  - SC Grand Med SRL, Oradea, Bihor County
  - S.C. Endodigest S.R.L., Oradea, Bihor County
  - SC Ames Research Center SRL, Clarasi, Calaras
  - S.C. Centrul Medical Unirea S.R.L., Cluj-Napoca, Cluj
  - S.C. Top Diabet Srl, Craiova, Dolj
  - County Hospital Deva, Deva, Hunedoara County
  - CMI Dr Pop Lavinia, Baia Mare, Maramureş
  - Sc Mediab Srl, Târgu Mureş, Mureș County
  - 3rd Clinic for Nutrition-Spitalulul Județean de Urgenta, Timișoara, Timiș County
  - Minimed S.R.L., Bacau
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed, Brasov
  - Sc Nicodiab Srl, Bucharest
  - "Carol Davila" Military Emergency Hospital, Bucharest
  - Sana Monitoring SRL, Bucharest
  - Institutul National de Endocrinologie C.I. Parhon, Bucharest
  - SC Eco-Diagnosis SRL, Bucharest
  - S.C. Medcon S.R.L, Buzău
  - S.C Milena Sante SRL, Galati
  - SC Diamed Obesity SRL, Galati
  - SC Consultmed SRL, Iași
  - SC Cardiomed SRL, Iași
  - Centrul Medical Bella Praxis, Paşcani
  - Bella Praxis S.R.L., Paşcani
  - S.C. Dianutrilife Medica S.R.L., Ploieşti
  - County Emergency Hospital Satu Mare, Satu Mare
  - SC Gensan SRL, Policlinica ASTRA, Sibiu
- Russia (49):
  - Tumen State Medical University, Tyumen, Russia
  - Volosevich First City Clinical Hospital, Arkhangelsk
  - Reg. State Budget Healthc. Inst. Regional Clinical Hospital, Barnaul
  - City Hospital #5, Barnaul
  - RBSHI "Altay Regional Cardiology Dispensary", Barnaul
  - Belgorod regional clinical hospital of the St. Ioasaph, Belgorod
  - Cardiological dispensary, Ivanovo
  - KSFMU, Inrereginal Clinical Diagnostic center, Kazan'
  - Institute of Complex Problems of Cardio-Vascular Diseases, Kemerovo
  - Medical Center CAPITAL-HEALTH, Moscow
  - Moscow City Clinical Hospital #15, Moscow
  - Friendship University of Russia, Moscow
  - Moscow State University n.a. M.V. Lomonosov, Moscow
  - National Medical Research Center of Cardiology, Moscow
  - City Clinical Hospital №52, Moscow
  - Federal Bureau for Medical and Social Expertise, Moscow
  - PHI "Central Clinical Hospital RZD- Medicine", Moscow
  - Moscow City Clinical Hospital n.a. A.K. Eramishantseva, Moscow
  - LLC RC Medical, Novosibirsk
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - LLC Reafan, Novosibirsk
  - Scientific Research Institute of neuroscience and Medicine, Novosibirsk
  - Orenburg Regional Clinical Hospital, Orenburg
  - Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - Rostov State Medical University_Rostov-on-Don, Rostov-on-Don
  - City policlinic #28, Saint Petersburg
  - Joint Stock Company "Modern Medical Technologies", Saint Petersburg
  - SPb SBHI City Outpatient clinic #37, Saint Petersburg
  - SPb SBHI City Outpatient clinic #109, Saint Petersburg
  - Limited Liability Company "Energiya Zdoroviya", Saint Petersburg
  - SPb SBHI City Multifield Hospital #2, Saint Petersburg
  - SPb SBHI City polyclinic #117, Saint Petersburg
  - FSPbSMU n.a. Academic I.P. Pavlov, Saint Petersburg
  - Consultative & Diagnostic Center with a Outpatient Hospital, Saint Petersburg
  - Saint-Petersburg "City Policlinic # 74", Saint Petersburg
  - Astarta Clinic LLC, Saint Petersburg
  - SPb SBHI City Hospital #38 n.a. N.A. Semashko, Saint-Petersburg, Pushkin
  - Regional Clinical cardiological dispensary n.a. Polyakov, Samara
  - City Hospital #4, Sochi, Sochi
  - SAHI of Komi Republic "Consultative Diagnostic Center", Syktyvkar
  - Tomsk National Research Medical Center of the RAS, Tomsk
  - Tomsk Regional Clinical Hospital, Tomsk
  - Siberian State Medical University_Tomsk, Tomsk
  - Regional Clinical Hospital of Tver, Tver'
  - Tumen State Medical University - RIMBB, Tyumen
  - Ulianovsk Regional Clinical Hospital, Ulyanovsk
  - Voronezh Regional Clinical Consultive-diagnostic Centre, Voronezh
  - Solovyov Clinical Emergency Hospital, Yaroslavl
  - Urals State Medical University, Yekaterinburg
- Serbia (6):
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad, Vojvodina
  - Clinical centre of Serbia, Clinic for cardiology, Belgrade
  - Clinical Centre of Serbia, Emergency Centre, Department of Cardiology, Belgrade
  - Emergency Internal Medicine Clinic, Belgrade
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Special Hospital "Sveti Sava", Belgrade
- South Africa (25):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Cardiology Research_Bloemfontein, Bloemfontein, Free State
  - IATROS International, Bloemfontein, Free State
  - Josha Research, Bloemfontein, Free State
  - Cardiology Clinical Research, Alberton, Gauteng
  - Dr Iftikhar Osman Ebrahim, Centurion, Gauteng
  - CRISMO, Germiston, Gauteng
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Tickerdoc Research (Pty) LTD, Johannesburg, Gauteng
  - WITS Clinical Research, Johannesburg, Gauteng
  - Dr Moosa's Rooms, Lenasia, Gauteng
  - Lenasia Clinical Trial Centre, Lenasia, Gauteng
  - Jongaie Research, Pretoria, Gauteng
  - Synexus Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Clinical Trial Systems (CTC), Pretoria, Gauteng
  - Roodepoort Medicross Clinical Research Centre, Roodepoort, Gauteng
  - Dr Jugnundan's Rooms, Durban, KwaZulu-Natal
  - Dr S Dawood, Cape Town, Western Cape
  - Dr Corbett, Cape Town, Western Cape
  - Tread Research (Pty)Ltd, Cape Town, Western Cape
  - UCT Lung institute, Cape Town, Western Cape
  - Cape Town Medical Research Centre, Kuilsriver, Western Cape
  - Paarl Research Centre, Paarl, Western Cape
  - Synexus Helderberg Clinical Research Centre, Somerset West, Western Cape
  - Clinical Projects Research, Worcester, Western Cape
- Spain (11):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Periférico de Especialidades Bola Azul, Almería
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Virgen de la Victoria, Málaga
  - Hospital Son Llatzer, Palma de Mallorca
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Virgen de la Macarena, Seville
  - Hospital Infanta Luisa, Seville
  - Hospital La Fe - Endocrinología y Nutrición, Valencia
- Sweden (6):
  - Lundberglab for Diab Research, Gothenburg
  - Centralsjukhuset, Kristianstad, Kristianstad
  - Clemenstorgets Hjärtmottagning, Lund
  - Enheten för Kliniska Studier (EKS), Örebro, Örebro
  - Hjärtenheten, Östersund
  - Karolinska Universitetssjukhuset Solna,FOU Tema Hjärta Kärl, Stockholm
- Taiwan (5):
  - HsinChu MacKay Memorial Hospital, Hsinchu
  - E-DA Hosiptal, Kaohsiung City
  - MacKay Memorial Hospital-Tamsui Branch, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan
- Thailand (9):
  - Thammasat University Hospital, Klong Luang, Pathumthani, Changwat Pathum Thani
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Mueang Chiang Mai District
  - King Chulalongkorn Memorial Hospital_Bangkok, Bangkok
  - Phramongkutklao Hospital-cardio, Bangkok
  - Phramongkutklao Hospital-neuro, Bangkok
  - Ramathibodi Hospital-Cardiovascular metabolic Center, Bangkok
  - Siriraj Hospital_Bangkok_1, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital-cardio, Chiang Mai
  - Srinakarind Hospital-Division of Cardiology, Khon Kaen
- Turkey (Türkiye) (21):
  - Baskent Universitesi Adana, Adana
  - Cukurova University School of Medicine Balcali Hospital, Adana
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Akdeniz University Tip Fakultesi Hastanesi, Antalya
  - Adnan Menderes Universitesi Uygulama ve Arastirma Hastanesi, Aydin
  - Eskisehir Osmangazi University-Cardio, Eskişehir
  - Gaziantep Universitesi Tip Fakultesi Hastanesi, Gaziantep
  - Koc University Hospital, Istanbul
  - Seyrantepe Hamidiye Etfal Egitim ve Arastirma Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi - Endokrinoloji, Istanbul
  - TC SB Ist.İl Sag.Müd.Prof.Dr.Cemil Tascioglu Sehir Hastanesi, Istanbul
  - Fatih Sultan Mehmet Hastanesi, Istanbul
  - Umraniye Egitim ve Arastirma Hastanesi, Istanbul
  - T.C. Saglik Bakanligi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Ege University School of Medicine, Cardiology Department, Izmir
  - Izmir Tepecik Training and Research Hospital, Izmir
  - Dokuz Eylul University School of Medicine, Cardiology, Izmir
  - Erciyes University Cardiology, Kayseri
  - Mersin University Cardiology, Mersin
  - Cumhuriyet University School of Medicine-Cardiology, Sivas
- Ukraine (17):
  - CMI City Clinical Hospital #3, Chernivtsi
  - CNPI "Kharkiv City Clinical Hospital #27", Kharkiv
  - NI of Therapy na LT Malaya of NAMSU - Chr. Non-Communicable, Kharkiv
  - Oleksandrivska Clinical Hospital - cardio rehabilitation dep, Kyiv
  - Medical Center of LLC 'Harmoniya Krasy', Kyiv
  - Medical Center 'Ok!Clinic+' of II of Clinical Studies LLC, Kyiv
  - Kyiv City Clinical Hospital of Emergency Care - Infarction, Kyiv
  - Clinical Hosp on the railway line №2 branch PHC JSC Ukrzaliz, Kyiv
  - MD Strazheska Institute of Cardiology of NAMSU - Resuscitati, Kyiv
  - Kyiv Regional Hospital, Kyiv
  - City Clinical Emergency Hospital - Cardiology department, Lviv
  - Odesa Regional Clinical Hospital, Odesa
  - Odessa Clinical Railway Hospital - Outpatient department, Odesa
  - City Clinical Hospital #1 - Therapy department, Vinnytsia
  - Vinnytsia Regional Clinical Hospital - Cardiology department, Vinnytsia
  - Central City Hospital #1 - Scientific-Research center, Zhytomyr
  - Zhytomir Regional Clinical Hospital - Cardio-Arrhytm. centre, Zhytomyr
- United Kingdom (42):
  - Harrogate District Hospital, Harrogate, North Yorkshire
  - Clifton Medical Centre, Rotherham, South Yorkshire
  - St. Richards Hospital, Chichester, West Sussex
  - Crouch Oak Family Practice, Addlestone
  - Stroke Trials Office, Airdrie
  - Antrim Area Hospital, Antrim
  - Axbridge & Wedmore Medical Practice, Axbridge
  - Bermuda Practice, Basingstoke
  - Sea Road Surgery, Bexhill-on-Sea
  - Birmingham Heartlands Hospital, Birmingham
  - Layton Medical Centre, Blackpool
  - Bollington Medical Centre, Bollington
  - The Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - Ely Bridge Surgery, Cardiff
  - St Peters Hospital, Chertsey, Chertsey
  - Countess Of Chester NHS Foundation Trust, Chester
  - WISDEM Centre, Coventry
  - Ninewells Hospital, Dundee
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Department Of Cardiac Research, Harrow
  - Wycombe General Hospital, High Wycombe
  - Hull Royal Infirmary, Hull
  - Cardiology, Leicester
  - Lincoln County Hospital, Lincoln
  - University Hospital Aintree, Liverpool
  - Guys Hospital, London
  - Kings College Hospital, London
  - Imperial College London, London
  - Diabetes Centre North Manchester General Hospital, Manchester
  - Cardio Research, Middlesbrough
  - University Dept of Medicine, Derriford Hospital, Plymouth, Plymouth
  - Clarence Medical Centre, Rhyl
  - Ashfields Primary Care Centre, Sandbach
  - Clinical Research Unit, Somerset
  - Moorgreen Hospital, Southampton
  - Lister Hospital, Stevenage
  - Sunderland Royal Hospital, Sunderland
  - Musgrove Park Hospital, Taunton
  - Cardiology Department, Torquay
  - Royal Cornwall Hospital (Treliske), Truro
  - University Hospital Wishaw, Wishaw

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Ryan DH, Lingvay I, Colhoun HM, Deanfield J, Emerson SS, Kahn SE, Kushner RF, Marso S, Plutzky J, Brown-Frandsen K, Gronning MOL, Hovingh GK, Holst AG, Ravn H, Lincoff AM. Semaglutide Effects on Cardiovascular Outcomes in People With Overweight or Obesity (SELECT) rationale and design. Am Heart J. 2020 Nov;229:61-69. doi: 10.1016/j.ahj.2020.07.008. Epub 2020 Jul 17. PMID 32916609
- [Result] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Result] Lincoff AM, Brown-Frandsen K, Colhoun HM, Deanfield J, Emerson SS, Esbjerg S, Hardt-Lindberg S, Hovingh GK, Kahn SE, Kushner RF, Lingvay I, Oral TK, Michelsen MM, Plutzky J, Tornoe CW, Ryan DH; SELECT Trial Investigators. Semaglutide and Cardiovascular Outcomes in Obesity without Diabetes. N Engl J Med. 2023 Dec 14;389(24):2221-2232. doi: 10.1056/NEJMoa2307563. Epub 2023 Nov 11. PMID 37952131
- [Derived] Nicholls SJ, Ryan DH, Deanfield J, Ferreira D, Lang CC, Lincoff AM, Lingvay I, Lubker C, Terns PP, Rasmussen S, Stensen S, Weeke PE, Kahn SE; SELECT Trial Investigators. Semaglutide and Hospitalizations in Patients With Obesity and Established Cardiovascular Disease: An Exploratory Analysis of the SELECT Randomized Clinical Trial. JAMA Cardiol. 2025 Dec 23:e254824. doi: 10.1001/jamacardio.2025.4824. Online ahead of print. PMID 41433034
- [Derived] Deanfield J, Lincoff AM, Kahn SE, Emerson SS, Lingvay I, Scirica BM, Plutzky J, Kushner RF, Colhoun HM, Hovingh GK, Stensen S, Weeke PE, Jeppesen OK, Bravo R, Wu CC, Komuro I, Santini F, Hjelmesaeth J, Urina-Triana M, Buscemi S, Ryan DH. Semaglutide and cardiovascular outcomes by baseline and changes in adiposity measurements: a prespecified analysis of the SELECT trial. Lancet. 2025 Nov 8;406(10516):2257-2268. doi: 10.1016/S0140-6736(25)01375-3. Epub 2025 Oct 22. PMID 41138739
- [Derived] Lubker C, Bhavsar J, Duque do Vale R, Emerson SS, Nortoft E, Plutzky J, Roberts G, Tarp JM, Lincoff AM. The Composite Number Needed to Treat for Semaglutide in Populations with Overweight or Obesity and Established Cardiovascular Disease Without Diabetes. Adv Ther. 2025 May;42(5):2513-2525. doi: 10.1007/s12325-025-03176-w. Epub 2025 Mar 29. PMID 40156748
- [Derived] McEwan P, Bog M, Faurby M, Foos V, Lingvay I, Lubker C, Miller R, Toliver JC, Yeates F, Lincoff AM. Cost-effectiveness of semaglutide in people with obesity and cardiovascular disease without diabetes. J Med Econ. 2025 Dec;28(1):268-278. doi: 10.1080/13696998.2025.2459529. Epub 2025 Feb 12. PMID 39882599
- [Derived] Badve SV, Bilal A, Lee MMY, Sattar N, Gerstein HC, Ruff CT, McMurray JJV, Rossing P, Bakris G, Mahaffey KW, Mann JFE, Colhoun HM, Tuttle KR, Pratley RE, Perkovic V. Effects of GLP-1 receptor agonists on kidney and cardiovascular disease outcomes: a meta-analysis of randomised controlled trials. Lancet Diabetes Endocrinol. 2025 Jan;13(1):15-28. doi: 10.1016/S2213-8587(24)00271-7. Epub 2024 Nov 25. PMID 39608381
- [Derived] Mendonca L, Moura H, Chaves PC, Neves JS, Ferreira JP. The Impact of Glucagon-Like Peptide-1 Receptor Agonists on Kidney Outcomes: A Meta-Analysis of Randomized Placebo-Controlled Trials. Clin J Am Soc Nephrol. 2024 Oct 8;20(2):159-68. doi: 10.2215/CJN.0000000584. Online ahead of print. PMID 39480988
- [Derived] Kosiborod MN, Deanfield J, Pratley R, Borlaug BA, Butler J, Davies MJ, Emerson SS, Kahn SE, Kitzman DW, Lingvay I, Mahaffey KW, Petrie MC, Plutzky J, Rasmussen S, Ronnback C, Shah SJ, Verma S, Weeke PE, Lincoff AM; SELECT, FLOW, STEP-HFpEF, and STEP-HFpEF DM Trial Committees and Investigators. Semaglutide versus placebo in patients with heart failure and mildly reduced or preserved ejection fraction: a pooled analysis of the SELECT, FLOW, STEP-HFpEF, and STEP-HFpEF DM randomised trials. Lancet. 2024 Sep 7;404(10456):949-961. doi: 10.1016/S0140-6736(24)01643-X. Epub 2024 Aug 30. PMID 39222642
- [Derived] Scirica BM, Lincoff AM, Lingvay I, Bogdanski P, Buscemi S, Colhoun H, Craciun AE, Ezhov M, Hardt-Lindberg S, Kleist Jeppesen O, Matos ALSA, Node K, Schiele F, Toplak H, van Beek A, Weeke PE, Wiviott SD, Deanfield J, Ryan D. The Effect of Semaglutide on Mortality and COVID-19-Related Deaths: An Analysis From the SELECT Trial. J Am Coll Cardiol. 2024 Oct 22;84(17):1632-1642. doi: 10.1016/j.jacc.2024.08.007. Epub 2024 Aug 30. PMID 39217559
- [Derived] Deanfield J, Verma S, Scirica BM, Kahn SE, Emerson SS, Ryan D, Lingvay I, Colhoun HM, Plutzky J, Kosiborod MN, Hovingh GK, Hardt-Lindberg S, Frenkel O, Weeke PE, Rasmussen S, Goudev A, Lang CC, Urina-Triana M, Pietila M, Lincoff AM; SELECT Trial Investigators. Semaglutide and cardiovascular outcomes in patients with obesity and prevalent heart failure: a prespecified analysis of the SELECT trial. Lancet. 2024 Aug 24;404(10454):773-786. doi: 10.1016/S0140-6736(24)01498-3. PMID 39181597
- [Derived] Colhoun HM, Lingvay I, Brown PM, Deanfield J, Brown-Frandsen K, Kahn SE, Plutzky J, Node K, Parkhomenko A, Ryden L, Wilding JPH, Mann JFE, Tuttle KR, Idorn T, Rathor N, Lincoff AM. Long-term kidney outcomes of semaglutide in obesity and cardiovascular disease in the SELECT trial. Nat Med. 2024 Jul;30(7):2058-2066. doi: 10.1038/s41591-024-03015-5. Epub 2024 May 25. PMID 38796653
- [Derived] Ryan DH, Lingvay I, Deanfield J, Kahn SE, Barros E, Burguera B, Colhoun HM, Cercato C, Dicker D, Horn DB, Hovingh GK, Jeppesen OK, Kokkinos A, Lincoff AM, Meyhofer SM, Oral TK, Plutzky J, van Beek AP, Wilding JPH, Kushner RF. Long-term weight loss effects of semaglutide in obesity without diabetes in the SELECT trial. Nat Med. 2024 Jul;30(7):2049-2057. doi: 10.1038/s41591-024-02996-7. Epub 2024 May 13. PMID 38740993
- [Derived] Rowe IA, Allen AM. Hepatic steatosis provides the terroir that promotes the development of cardiovascular risk factors and disease. Hepatology. 2023 Jun 1;77(6):1843-1845. doi: 10.1097/HEP.0000000000000327. Epub 2023 Feb 6. No abstract available. PMID 36738088
- [Derived] Leite AR, Angelico-Goncalves A, Vasques-Novoa F, Borges-Canha M, Leite-Moreira A, Neves JS, Ferreira JP. Effect of glucagon-like peptide-1 receptor agonists on cardiovascular events in overweight or obese adults without diabetes: A meta-analysis of placebo-controlled randomized trials. Diabetes Obes Metab. 2022 Aug;24(8):1676-1680. doi: 10.1111/dom.14707. Epub 2022 May 3. PMID 35373878
- [Derived] Mares AC, Chatterjee S, Mukherjee D. Semaglutide for weight loss and cardiometabolic risk reduction in overweight/obesity. Curr Opin Cardiol. 2022 Jul 1;37(4):350-355. doi: 10.1097/HCO.0000000000000955. Epub 2022 Feb 16. PMID 35175229
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were screened at 811 sites in 41 countries. Out of 811 sites, participants were randomised at 804 sites.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive treatment with either semaglutide or placebo as an adjunct to standard-of-care.
Groups:
- Semaglutide: Participants received semaglutide subcutaneously once weekly in a fixed-dose escalation manner, with dose increases every 4 weeks for up to week 16 (0.25 milligrams [mg], 0.5 mg, 1.0 mg and 1.7 mg) followed by maintenance dose of 2.4 mg once weekly up to the end of treatment period.
- Placebo: Participants received placebo (matched to semaglutide) subcutaneously once weekly up to the end of treatment period.
Period: Overall Study
Arm/Group | Semaglutide | Placebo
Started | 8803 | 8801
Full Analysis Set (FAS) (FAS included all randomised participants. All participants were analyzed according to the treatment to which they were assigned at randomisation.) | 8803 | 8801
Completed (Participants attended follow-up visit or died during trial considered completers in the trial.) | 8544 | 8517
Not Completed | 259 | 284
Not completed — Withdrawal by Subject | 67 | 96
Not completed — Lost to Follow-up | 192 | 188

BASELINE CHARACTERISTICS:
Population: FAS included all randomised participants. All participants were analyzed according to the treatment to which they were assigned at randomisation.
Groups:
- Semaglutide: Participants received semaglutide subcutaneously once weekly in a fixed-dose escalation manner, with dose increases every 4 weeks for up to week 16 (0.25 mg, 0.5 mg, 1.0 mg and 1.7 mg) followed by maintenance dose of 2.4 mg once weekly up to the end of treatment period.
- Total: Total of all reporting groups
Arm/Group | Semaglutide | Placebo | Total
Number analyzed (Participants) | 8803 | 8801 | 17604
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (8.9) | 61.6 (8.8) | 61.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2448 | 2424 | 4872
  Male | 6355 | 6377 | 12732
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 914 | 908 | 1822
  Not Hispanic or Latino | 7794 | 7817 | 15611
  Unknown or Not Reported | 95 | 76 | 171
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 23 | 21 | 44
  Asian | 720 | 727 | 1447
  Black or African American | 348 | 323 | 671
  Native Hawaiian or Other Pacific Islander | 3 | 5 | 8
  White | 7387 | 7404 | 14791
  Other | 227 | 247 | 474
  Not Reported | 95 | 74 | 169

OUTCOME MEASURES:

1. Primary Outcome: Participants From Time of Randomization to First Occurrence of a Composite Outcome Measure Consisting of: Cardiovascular (CV) Death, Non-fatal Myocardial Infarction (MI), or Non-fatal Stroke
Description: Number of participants with first occurrence of composite outcome measure consisted of CV death (undetermined cause of death presumed CV death), non-fatal MI, or non-fatal stroke are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 569 | 701
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Data from the in-trial period. The outcome measure was analysed using a Cox proportional hazards model with treatment as categorical fixed factor. Participants without events of interest were censored at the end of their in-trial period; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.72 to 0.89]

2. Secondary Outcome: Participants From Time of Randomisation to CV Death
Description: Number of participants with CV death are presented. The outcome measure was evalulated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 223 | 262

3. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of a Composite Heart Failure (HF) Outcome Measure Consisting of: HF Hospitalisation, Urgent HF Visit or CV Death
Description: Number of participants with first occurrence of a composite HF outcome measure consisted of HF hospitalisation, urgent HF visit or CV death are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 300 | 361

4. Secondary Outcome: Participants From Time of Randomisation to All-cause Death
Description: Number of participants with all-cause death are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 375 | 458

5. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of an Expanded Composite CV Outcome Measure Consisting of: CV Death, Non-fatal MI, Non-fatal Stroke, Coronary Revascularisation or Unstable Angina Pectoris (UAP) Requiring Hospitalisation
Description: Number of participants with first occurrence of an expanded composite CV outcome measure consisted of CV death, non-fatal MI, non-fatal stroke, coronary revascularisation or UAP requiring hospitalisation are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 873 | 1074

6. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of a Composite Outcome Measure Consisting of: All-cause Death, Non-fatal MI, or Non-fatal Stroke
Description: Number of participants with first occurrence of a composite outcome measure consisted of all-cause death, non-fatal MI, or non-fatal stroke are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 710 | 877

7. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of Non-fatal MI
Description: Number of participants with first occurrence of non-fatal MI are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 234 | 322

8. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of Non-fatal Stroke
Description: Number of participants with first occurrence of non-fatal stroke are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 154 | 165

9. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of Coronary Revascularisation
Description: Number of participants with first occurrence of coronary revascularisation are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 473 | 608

10. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of UAP Requiring Hospitalisation
Description: Number of participants with first occurrence of UAP requiring hospitalisation are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 109 | 124

11. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of HF Requiring Hospitalisation or Urgent HF Visit
Description: Number of participants with first occurrence of HF requiring hospitalisation or urgent HF visit are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 97 | 122

12. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of Glycosylated Haemoglobin (HbA1c) Greater Than Equals to (≥) 48 Millimole Per Mole (mmol/Mol) (6.5 Percentage [%])
Description: Number of participants with first occurrence of HbA1c ≥ 48 mmol/mol (6.5%) are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: FAS included all randomised participants. All participants were analyzed according to the treatment to which they were assigned at randomisation. Here, overall number of participants analyzed = number of participants with HbA1c less than (<) 48 mmol/mol (6.5%) at screening. Participants with ≥ 48 mmol/mol (6.5%) at screening were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8800 | 8797
Participants | 306 | 1059

13. Secondary Outcome: Participants From Time of Randomisation to First Occurrence of a 5-component Composite Nephropathy Outcome Measure
Description: Number of participants with first occurrence of a 5-component composite nephropathy outcome measure consisted of onset of persistent macroalbuminuria (UACR > 300 milligram per gram [mg/g]), persistent 50% reduction in estimated glomerular filtration rate (eGFR) compared with baseline (randomisation), onset of persistent eGFR < 15 ml/min/1.73m^2, initiation of chronic renal replacement therapy (dialysis or transplantation) or renal death. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 8803 | 8801
Participants | 155 | 198

14. Secondary Outcome: Participants From Time of Randomisation to HbA1c ≥ 39 mmol/Mol (5.7%) (for Participants With a Screening HbA1c <39 mmol/Mol [5.7%])
Description: Number of participants with HbA1c ≥ 39 mmol/mol (5.7%) are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: From randomisation (week 0) up to 240 weeks
Population: FAS included all randomised participants. All participants were analyzed according to the treatment to which they were assigned at randomisation. Here, overall number of participants analyzed = number of participants with HbA1c <39 mmol/mol (5.7%) at screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 2925 | 2980
Participants | 623 | 1501

15. Secondary Outcome: Participants With HbA1c < 39 mmol/Mol (5.7%) (for Participants With a Screening HbA1c ≥ 39 mmol/Mol [5.7%])
Description: Number of participants with HbA1c < 39 mmol/mol (5.7%) are presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: At week 52, week 104
Population: FAS included all randomised participants. All participants were analyzed according to the treatment to which they were assigned at randomisation. Here, overall number of participants analyzed = number of participants with HbA1c ≥ 39 mmol/mol (5.7%) at screening. And, number analyzed = number of participants who contributed to the analysis at that particular timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 5877 | 5819
Participants
  Week 52: number analyzed (Participants) | 5112 | 5078
  Week 52 | 3363 | 955
  Week 104: number analyzed (Participants) | 4971 | 4864
  Week 104 | 3271 | 978

16. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change in SBP from randomisation (week 0) to week 104 is presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: FAS included all randomised participants. All participants were analyzed according to the treatment to which they were assigned at randomisation. Here, overall number of participants analyzed = number of participants who contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Millimetre of mercury (mmHg)
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7475 | 7385
Millimetre of mercury (mmHg) | -3.8 (16.4) | -0.6 (16.0)

17. Secondary Outcome: Change in Diastolic Blood Pressure (DBP)
Description: Change in DBP from randomisation (week 0) to week 104 is presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7475 | 7384
mmHg | -1.1 (10.4) | -0.4 (10.4)

18. Secondary Outcome: Change in Pulse
Description: Change in pulse from randomisation (week 0) to week 104 is presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: beats per mintue (bpm)
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7473 | 7385
beats per mintue (bpm) | 3.8 (11.0) | 0.9 (10.7)

19. Secondary Outcome: Change in High Sensitivity C-Reactive Protein (hsCRP) - Ratio to Baseline
Description: Change in hsCRP (milligram per liter [mg/L]) from randomisation (week 0) to week 104 presented as ratio to baseline (week 0). The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of hsCRP
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7472 | 7400
ratio of hsCRP | 0.61 (149.53) | 1.00 (133.25)

20. Secondary Outcome: Change in Total Cholesterol - Ratio to Baseline
Description: Change in total cholesterol (milligram per deciliter [mg/dL]) from randomisation (week 0) to week 104 is presented as ratio to baseline (week 0). The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of total cholesterol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7461 | 7394
ratio of total cholesterol | 0.95 (21.54) | 0.98 (21.24)

21. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol - Ratio to Baseline
Description: Change in HDL (mg/dL) from randomisation (week 0) to week 104 is presented as ratio to baseline (week 0). The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of HDL
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7137 | 7091
ratio of HDL | 1.05 (17.39) | 1.01 (16.69)

22. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol - Ratio to Baseline
Description: Change in LDL (mg/dL) from randomisation (week 0) to week 104 is presented as ratio to baseline (week 0). The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of LDL
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7138 | 7088
ratio of LDL | 0.95 (37.43) | 0.97 (37.83)

23. Secondary Outcome: Change in Triglycerides - Ratio to Baseline
Description: Change in triglycerides (mg/dL) from randomisation (week 0) to week 104 is presented as ratio to baseline (week 0). The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of triglycerides
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7432 | 7364
ratio of triglycerides | 0.82 (46.33) | 0.97 (44.31)

24. Secondary Outcome: Change in Body Weight
Description: Percentage change in body weight from randomisation (week 0) to week 104 is presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percentage change in body weight
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7474 | 7378
percentage change in body weight | -9.39 (8.62) | -0.87 (6.08)

25. Secondary Outcome: Change in Waist Circumference
Description: Change is waist circumference from randomisation (week 0) to week 104 is presented. The outcome measure was evaluated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7373 | 7273
centimeter (cm) | -7.5 (9.4) | -1.0 (7.3)

26. Secondary Outcome: Change From Randomisation (Week 0) in Participant Reported Outcome (PRO): EuroQol Five Dimensions Five Level Questionnaire (EQ-5D-5L) Index Score to Week 104
Description: EQ-5D-5L is a PRO tool used to estimate impact on participant's health-related quality of life and provides a description of their problems by dimensions (descriptive system). EQ-5D has 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression, and each dimension has 5 levels: not at all, mild, moderate, severe, extreme. Participant marks most appropriate statement in each dimension, resulting in 1-digit number and digits from 5 dimensions can be combined in 5-digit number describing participant's health state. Index score records an average health status according to dimensions using an algorithm, ranges 0-1 with higher score indicates better health status. Outcome measure was evaluated based on data from in-trial observation period (defined as date of randomisation to one of the dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant [who were lost to follow-up], date of death).
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 6761 | 6665
score on a scale | 0.01 (0.14) | -0.01 (0.14)

27. Secondary Outcome: Change From Randomisation (Week 0) in PRO: EuroQol Five Dimensions Visual Analogue Scale (EQ-5D-VAS) to Week 104
Description: EQ-5D-5L is a PRO tool used to estimate impact on participant's health-related quality of life and provides a description of their problems by dimensions (descriptive system). EQ-5D has 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression, and each dimension has 5 levels: not at all, mild, moderate, severe, extreme. Participant marks most appropriate statement in each dimension, resulting in 1-digit number and digits from 5 dimensions can be combined in 5-digit number describing participant's health state. VAS component records a participant's overall self-rated health on a range of 0-100 with higher score indicates better self-reported health status. Outcome measure was evaluated based on data from in-trial observation period (defined as date of randomisation to one of the dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant [who were lost to follow-up], date of death).
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 6761 | 6665
score on a scale | 2.38 (15.38) | 0.77 (15.79)

28. Secondary Outcome: Change in HbA1c - Percentage
Description: Change in HbA1c (percentage) from randomisation (week 0) to week 104 is presented. The outcome measure was evaulated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7439 | 7351
Percentage of HbA1c | -0.31 (0.37) | 0.01 (0.36)

29. Secondary Outcome: Change in HbA1c - mmol/Mol
Description: Change in HbA1c (mmol/mol) from randomisation (week 0) to week 104 is presented. The outcome measure was evaulated based on data from in-trial observation period. In-trial observation period defined as the period from date of randomisation to one of the following dates, whichever comes first: date of follow-up visit, date when participant withdrew consent, date of last contact with participant for participants who were lost to follow-up (participant did not complete the trial and did not withdraw consent), date of death.
Time Frame: Week 0, week 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 7439 | 7351
mmol/mol | -3.38 (4.06) | 0.10 (3.94)

ADVERSE EVENTS:
Time Frame: From randomisation (week 0) up to 240 weeks
Description: AEs are reported based on data from in-trial observation period. Not all the AEs were collected systematically and more details on the approach followed for collecting the AEs is mentioned in the section 9.2 of protocol. AEs were not separately collected for each dose level. Hence, AEs are presented in randomized arm (semaglutide vs placebo).
Arm/Group | Semaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 371/8803 | 460/8801
Serious Adverse Events (participants affected / at risk) | 2941/8803 | 3204/8801
Other Adverse Events (participants affected / at risk) | 3944/8803 | 2440/8801
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=8803) | Placebo (N=8801)
Abdominal adhesions (Gastrointestinal disorders) | 7 (8) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 5 (5) | 6 (6)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 18 (19)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 11 (12) | 12 (12)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal symptom (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 3 (3)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 2 (2) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accident at home (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accident at work (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Accidental death (General disorders) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 22 (23) | 18 (18)
Acute kidney injury (Renal and urinary disorders) | 79 (87) | 105 (116)
Acute left ventricular failure (Cardiac disorders) | 6 (6) | 7 (8)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 209 (220) | 293 (324)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 28 (30) | 46 (51)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (16) | 15 (15)
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 4 (4)
Alcohol poisoning (Injury, poisoning and procedural complications) | 3 (3) | 3 (4)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 3 (3) | 2 (3)
Alcoholic liver disease (Hepatobiliary disorders) | 2 (2) | 0 (0)
Alcoholism (Psychiatric disorders) | 2 (2) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 5 (5)
Amylase increased (Investigations) | 2 (2) | 0 (0)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 36 (40) | 30 (38)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Anal abscess (Infections and infestations) | 5 (5) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 6 (6)
Anal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 4 (4)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 0 (0)
Aneurysm thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 116 (126) | 150 (176)
Angina unstable (Cardiac disorders) | 182 (205) | 209 (242)
Anginal equivalent (Cardiac disorders) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Angioplasty (Surgical and medical procedures) | 3 (3) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 5 (5) | 12 (12)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anorectal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anterior cord syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Anticoagulant-related nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 2 (2)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (8) | 3 (3)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 18 (18) | 17 (17)
Aortic aneurysm rupture (Vascular disorders) | 2 (2) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 4 (4) | 4 (4)
Aortic occlusion (Vascular disorders) | 0 (0) | 1 (1)
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 6 (6) | 19 (19)
Aortic valve incompetence (Cardiac disorders) | 3 (3) | 4 (4)
Aortic valve stenosis (Cardiac disorders) | 7 (8) | 6 (6)
Aorto-atrial fistula (Vascular disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 3 (3) | 3 (3)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 18 (18) | 16 (17)
Appendicitis perforated (Infections and infestations) | 6 (6) | 5 (5)
Appendix disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 7 (7) | 7 (7)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmic storm (Cardiac disorders) | 1 (1) | 1 (1)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial restenosis (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 7 (7) | 6 (6)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (19) | 11 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 10 (10)
Arthritis bacterial (Infections and infestations) | 1 (1) | 4 (4)
Arthritis infective (Infections and infestations) | 2 (2) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 10 (11) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 13 (18)
Ataxia (Nervous system disorders) | 1 (1) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 127 (139) | 152 (181)
Atrial flutter (Cardiac disorders) | 23 (24) | 22 (25)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial septal defect repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 6 (7)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 4 (4) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 7 (7) | 8 (9)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 4 (4) | 7 (7)
Atypical pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 26 (28)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 2 (3) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (21) | 27 (36)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 2 (2)
Basilar artery aneurysm (Nervous system disorders) | 3 (3) | 1 (1)
Basilar artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Behcet's syndrome (Vascular disorders) | 0 (0) | 1 (1)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Benign duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Benign neoplasm of cervix uteri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 34 (35) | 21 (21)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 16 (16) | 10 (10)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 8 (8)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 17 (18)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2)
Blood calcitonin increased (Investigations) | 2 (2) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 10 (10) | 9 (9)
Blood osmolarity decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 2 (2) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Bone deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (17) | 6 (6)
Bradycardia (Cardiac disorders) | 9 (9) | 9 (9)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 3 (3) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 3 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast fibrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 9 (9) | 15 (15)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 2 (2) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 1 (1)
Burn infection (Infections and infestations) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
CADASIL (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 124 (126) | 137 (137)
COVID-19 pneumonia (Infections and infestations) | 119 (119) | 148 (148)
Calculus bladder (Renal and urinary disorders) | 3 (3) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 7 (7) | 4 (4)
Campylobacter gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 26 (26) | 33 (33)
Cardiac death (General disorders) | 1 (1) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 88 (114) | 113 (127)
Cardiac failure acute (Cardiac disorders) | 32 (46) | 44 (50)
Cardiac failure chronic (Cardiac disorders) | 23 (24) | 28 (29)
Cardiac failure congestive (Cardiac disorders) | 31 (37) | 36 (51)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac perfusion defect (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 2 (2) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 11 (11) | 11 (11)
Cardiogenic shock (Cardiac disorders) | 6 (6) | 10 (10)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 5 (5)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 2 (2)
Carotid arterial embolus (Nervous system disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 3 (3) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 5 (5)
Carotid artery stenosis (Nervous system disorders) | 22 (23) | 24 (26)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 2 (2)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 12 (14) | 18 (22)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 29 (31) | 41 (43)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Central nervous system inflammation (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system vasculitis (Nervous system disorders) | 1 (1) | 0 (0)
Central pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 3 (3) | 4 (4)
Cerebellar ischaemia (Nervous system disorders) | 0 (0) | 4 (4)
Cerebellar stroke (Nervous system disorders) | 3 (3) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral circulatory failure (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 7 (7) | 8 (8)
Cerebral infarction (Nervous system disorders) | 17 (18) | 23 (25)
Cerebral ischaemia (Nervous system disorders) | 8 (8) | 6 (6)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 (0) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 35 (36) | 48 (50)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 2 (2) | 4 (4)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (9)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cervicitis (Infections and infestations) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 4 (4) | 7 (9)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Chest pain (General disorders) | 44 (45) | 47 (48)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 6 (6) | 4 (7)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis infective (Infections and infestations) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 13 (13) | 15 (15)
Cholecystitis acute (Hepatobiliary disorders) | 27 (27) | 30 (31)
Cholecystitis chronic (Hepatobiliary disorders) | 10 (10) | 4 (4)
Cholecystitis infective (Infections and infestations) | 4 (4) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 44 (46) | 31 (33)
Cholelithiasis migration (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 1 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Chronic coronary syndrome (Cardiac disorders) | 3 (3) | 5 (5)
Chronic gastritis (Gastrointestinal disorders) | 4 (4) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 7 (7) | 7 (7)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Chronic lymphocytic leukaemia stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 32 (43) | 50 (63)
Chronic sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Circulatory collapse (Vascular disorders) | 3 (3) | 3 (3)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 8 (8)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 4 (4) | 3 (3)
Coagulation time shortened (Investigations) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Cognitive disorder (Nervous system disorders) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 14 (15) | 10 (11)
Colitis ischaemic (Gastrointestinal disorders) | 9 (9) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 5 (5)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 4 (4)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Completed suicide (Psychiatric disorders) | 5 (5) | 2 (2)
Complicated appendicitis (Infections and infestations) | 0 (0) | 4 (4)
Complication associated with device (General disorders) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Confusional state (Psychiatric disorders) | 4 (4) | 5 (5)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 6 (6)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Conus medullaris syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Corneal degeneration (Eye disorders) | 0 (0) | 1 (1)
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 (3) | 1 (1)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 48 (51) | 64 (68)
Coronary arterial stent insertion (Surgical and medical procedures) | 245 (270) | 279 (343)
Coronary artery bypass (Surgical and medical procedures) | 69 (69) | 79 (79)
Coronary artery disease (Cardiac disorders) | 79 (80) | 106 (113)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 4 (4)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 11 (11) | 12 (12)
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 44 (49) | 53 (58)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Coronary revascularisation (Surgical and medical procedures) | 23 (27) | 37 (38)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 2 (2) | 3 (3)
Corticobasal degeneration (Nervous system disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Cranial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Crush injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Culture positive (Investigations) | 0 (0) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 5 (5) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Death (General disorders) | 55 (55) | 57 (57)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 13 (14) | 13 (13)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 19 (21) | 14 (14)
Delirium (Psychiatric disorders) | 1 (1) | 2 (3)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 3 (3) | 0 (0)
Dengue haemorrhagic fever (Infections and infestations) | 0 (0) | 1 (1)
Dental alveolar anomaly (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 13 (14) | 10 (10)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 3 (3) | 7 (7)
Device failure (Product Issues) | 0 (0) | 2 (2)
Device loosening (Product Issues) | 3 (3) | 1 (1)
Device malfunction (Product Issues) | 2 (2) | 4 (4)
Device occlusion (Product Issues) | 1 (1) | 1 (1)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 3 (3) | 3 (3)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 16 (17)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Diffuse large B-cell lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Diplegia (Nervous system disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Dissociative amnesia (Psychiatric disorders) | 1 (2) | 0 (0)
Dissociative identity disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 14 (17) | 23 (26)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 5 (5)
Diverticulum intestinal (Gastrointestinal disorders) | 7 (7) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (2) | 5 (6)
Dizziness (Nervous system disorders) | 10 (10) | 14 (14)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 3 (3)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 3 (3) | 2 (3)
Dry gangrene (Vascular disorders) | 1 (1) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 4 (4) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 7 (7)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenitis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dural arteriovenous fistula (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 2 (2) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 35 (36)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 4 (4) | 2 (2)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 1 (1)
Electrocution (General disorders) | 1 (1) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0)
Embolic stroke (Nervous system disorders) | 6 (6) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (3) | 5 (5)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 3 (3)
Endocarditis (Infections and infestations) | 4 (4) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endocrine ophthalmopathy (Eye disorders) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Enlarged uvula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epididymal disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 2 (2) | 1 (1)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 4 (4) | 9 (9)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epiretinal membrane (Eye disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 6 (6)
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 10 (11) | 13 (13)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Excessive skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Exercise electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extraskeletal ossification (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 2 (2) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (2)
Facial paralysis (Nervous system disorders) | 2 (2) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 1 (1)
Factor II mutation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 51 (55) | 35 (39)
False positive investigation result (Investigations) | 1 (1) | 0 (0)
Fat necrosis (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Femoral artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 11 (11) | 9 (9)
Femur fracture (Injury, poisoning and procedural complications) | 13 (13) | 11 (11)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Focal peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 2 (2)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 3 (3) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Frontotemporal dementia (Nervous system disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gallbladder necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 2 (2) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 4 (4) | 4 (4)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric pH decreased (Investigations) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric polyps (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 5 (5) | 9 (9)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric volvulus (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastritis (Gastrointestinal disorders) | 14 (14) | 13 (13)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 15 (16) | 11 (12)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 22 (22) | 15 (17)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal organ contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (13) | 13 (13)
Gastroparesis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 4 (4) | 2 (2)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 3 (3)
Giant cell arteritis (Vascular disorders) | 2 (2) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 7 (7) | 4 (4)
Gout (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Graft infection (Infections and infestations) | 0 (0) | 2 (2)
Granuloma (General disorders) | 1 (1) | 0 (0)
Graves' disease (Endocrine disorders) | 0 (0) | 1 (1)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haematoma (Vascular disorders) | 4 (4) | 4 (4)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 16 (17) | 11 (11)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 7 (7) | 12 (12)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 4 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Hanging (General disorders) | 0 (0) | 1 (1)
Head and neck cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 8 (8) | 10 (10)
Headache (Nervous system disorders) | 7 (8) | 11 (11)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Heart transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 3 (3) | 0 (0)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 4 (4) | 3 (3)
Hemiplegia (Nervous system disorders) | 1 (1) | 2 (2)
Hemiplegic migraine (Nervous system disorders) | 2 (2) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 4 (4)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic fibrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 5 (5)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 1 (1) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 4 (4)
Hiatus hernia (Gastrointestinal disorders) | 4 (4) | 6 (6)
Hip fracture (Injury, poisoning and procedural complications) | 11 (11) | 3 (3)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hormone receptor positive HER2 negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 7 (8) | 11 (11)
Hydrocele (Congenital, familial and genetic disorders) | 2 (2) | 3 (3)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hydrometra (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 6 (6) | 3 (3)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperaldosteronism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 7 (8)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Hyperparathyroidism primary (Endocrine disorders) | 2 (2) | 1 (1)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 27 (30) | 24 (24)
Hypertensive crisis (Vascular disorders) | 4 (5) | 13 (15)
Hypertensive emergency (Vascular disorders) | 2 (2) | 3 (3)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 3 (3)
Hypertensive urgency (Vascular disorders) | 5 (5) | 13 (16)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 7 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (25) | 18 (18)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Hypoparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 23 (24) | 25 (30)
Hypothermia (General disorders) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 3 (3)
IIIrd nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 2 (2)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Iliac artery disease (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 3 (3)
Iliac artery stenosis (Vascular disorders) | 2 (2) | 6 (6)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 4 (4) | 0 (0)
Impaired healing (General disorders) | 6 (6) | 5 (5)
Implant site infection (Infections and infestations) | 1 (1) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 2 (2)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Infected bite (Infections and infestations) | 2 (2) | 0 (0)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 (3) | 5 (5)
Inferior vena cava stenosis (Vascular disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 9 (9) | 8 (8)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 39 (41) | 24 (24)
Injection site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 6 (6) | 8 (8)
International normalised ratio increased (Investigations) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 16 (17) | 15 (15)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Intestinal gangrene (Infections and infestations) | 1 (1) | 0 (0)
Intestinal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 11 (11) | 8 (10)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-cerebral aneurysm operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 5 (6)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 6 (6)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 (8) | 7 (7)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 9 (9) | 2 (2)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 2 (2)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 79 (87) | 80 (84)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 6 (6) | 7 (8)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Joint injury (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Kidney fibrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Lacunar infarction (Nervous system disorders) | 6 (6) | 2 (2)
Lacunar stroke (Nervous system disorders) | 2 (2) | 3 (3)
Large cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Large intestine infection (Infections and infestations) | 4 (4) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 11 (11) | 9 (10)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 6 (6)
Left ventricular failure (Cardiac disorders) | 4 (4) | 6 (6)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Leptospirosis (Infections and infestations) | 1 (1) | 0 (0)
Leriche syndrome (Vascular disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukoplakia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 3 (3) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Liposarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Liposuction (Surgical and medical procedures) | 1 (1) | 0 (0)
Lisfranc fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 3 (3) | 3 (3)
Loss of consciousness (Nervous system disorders) | 5 (6) | 4 (5)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 7 (7)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 5 (6) | 5 (5)
Lower urinary tract symptoms (Renal and urinary disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 5 (5) | 4 (4)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 19 (20) | 15 (15)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Lumbosacral plexus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 8 (8)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Lung carcinoma cell type unspecified stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lyme disease (Infections and infestations) | 1 (1) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 2 (2) | 2 (2)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Macroangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 3 (3)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Macular rupture (Eye disorders) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Maisonneuve fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 2 (3) | 5 (5)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 9 (9)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of uterine adnexa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 6 (6) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Mania (Psychiatric disorders) | 2 (2) | 0 (0)
Mantle cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (2)
Medical device site ulcer (General disorders) | 1 (1) | 0 (0)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 2 (4) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 1 (1) | 0 (0)
Meningoradiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Meniscopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Mental disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 4 (4) | 5 (5)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mesenteric abscess (Infections and infestations) | 0 (0) | 1 (1)
Mesenteric artery embolism (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 5 (5) | 3 (3)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 2 (3)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 6 (6) | 3 (3)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 7 (7)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 3 (4)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 10 (10)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 2 (2)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 13 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 2 (2) | 0 (0)
Mycetoma mycotic (Infections and infestations) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 3 (3)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 35 (36) | 31 (32)
Myocardial injury (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 21 (21) | 31 (31)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopericarditis (Cardiac disorders) | 1 (1) | 1 (2)
Narcotic bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasopharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (12) | 8 (8)
Neck deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 25 (27) | 24 (30)
Nephropathy (Renal and urinary disorders) | 1 (2) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 2 (2) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgic amyotrophy (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Neuroendocrine breast tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine carcinoma of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 88 (96) | 103 (112)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 4 (4) | 7 (7)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1)
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 2 (2)
Oedema mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 6 (6)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 3 (3)
Oesophageal adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Oesophageal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 3 (3) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 2 (2) | 1 (1)
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 3 (3)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 15 (15) | 10 (11)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 84 (93) | 79 (86)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 4 (4) | 4 (4)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis externa candida (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Pain (General disorders) | 2 (2) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 9 (9)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 5 (5) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 9 (12) | 14 (15)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Parkinson's disease (Nervous system disorders) | 0 (0) | 3 (3)
Parkinsonian rest tremor (Nervous system disorders) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 3 (3) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 8 (8) | 5 (5)
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penetrating aortic ulcer (Vascular disorders) | 0 (0) | 2 (2)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (5)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Percutaneous coronary intervention (Surgical and medical procedures) | 70 (81) | 114 (124)
Perianal streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 5 (5) | 4 (4)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 3 (3) | 4 (4)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 37 (41) | 45 (58)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 9 (10) | 4 (4)
Peripheral artery occlusion (Vascular disorders) | 6 (7) | 9 (15)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 2 (3) | 5 (5)
Peripheral artery stenosis (Vascular disorders) | 8 (8) | 10 (13)
Peripheral artery thrombosis (Vascular disorders) | 4 (4) | 3 (4)
Peripheral embolism (Vascular disorders) | 0 (0) | 3 (3)
Peripheral ischaemia (Vascular disorders) | 4 (4) | 5 (5)
Peripheral nerve lesion (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 4 (4) | 7 (7)
Peripheral venous disease (Vascular disorders) | 1 (1) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 3 (3) | 5 (5)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Philadelphia positive chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (6)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 16 (16)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 89 (102) | 132 (146)
Pneumonia aspiration (Infections and infestations) | 4 (4) | 9 (9)
Pneumonia bacterial (Infections and infestations) | 5 (5) | 6 (6)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 2 (2) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Popliteal artery entrapment syndrome (Vascular disorders) | 0 (0) | 1 (1)
Portal hypertensive biliopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Portosplenomesenteric venous thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 2 (2) | 3 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 12 (12) | 7 (8)
Post procedural infection (Infections and infestations) | 2 (2) | 6 (6)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural sepsis (Infections and infestations) | 1 (1) | 4 (4)
Post procedural stroke (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post stroke epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Post stroke seizure (Nervous system disorders) | 1 (1) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 1 (1) | 2 (2)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Postoperative abscess (Infections and infestations) | 1 (1) | 3 (3)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Postoperative wound infection (Infections and infestations) | 8 (8) | 8 (8)
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 14 (14) | 15 (15)
Primary myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Primary progressive multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 3 (3) | 2 (2)
Procedural failure (General disorders) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 60 (60) | 54 (54)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 8 (8)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate infection (Infections and infestations) | 1 (1) | 1 (1)
Prostatic abscess (Infections and infestations) | 1 (1) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Prostatic obstruction (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Prostatomegaly (Reproductive system and breast disorders) | 5 (5) | 1 (1)
Prosthetic cardiac valve malfunction (Product Issues) | 0 (0) | 1 (1)
Prosthetic cardiac valve stenosis (General disorders) | 1 (1) | 1 (1)
Prosthetic valve endocarditis (Infections and infestations) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Pseudoaneurysm infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (2) | 1 (1)
Pseudoradicular syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Pseudostroke (Nervous system disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 38 (39) | 43 (44)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (12)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura fulminans (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 11 (11) | 7 (7)
Pyelonephritis acute (Infections and infestations) | 4 (4) | 2 (2)
Pyrexia (General disorders) | 5 (6) | 4 (6)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 5 (5)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 3 (3) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 2 (2)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Renal colic (Renal and urinary disorders) | 5 (5) | 1 (1)
Renal cortical necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 4 (4)
Renal impairment (Renal and urinary disorders) | 3 (3) | 6 (6)
Renal infarct (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal tubular dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal vein thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 16 (16)
Respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1)
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal artery thrombosis (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 5 (5) | 2 (2)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Retinal vascular occlusion (Eye disorders) | 2 (2) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reversible cerebral vasoconstriction syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 15 (16) | 21 (21)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 11 (11) | 17 (17)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 13 (15) | 5 (5)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 2 (2)
SARS-CoV-2 sepsis (Infections and infestations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 3 (3)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 2 (2) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Sciatic nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 7 (7) | 8 (9)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 1 (1)
Scrotal cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Scrotal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sebaceous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Secondary immunodeficiency (Immune system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 14 (14) | 6 (6)
Seizure like phenomena (Nervous system disorders) | 1 (1) | 2 (2)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (2)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 36 (36) | 35 (35)
Septic shock (Infections and infestations) | 11 (12) | 15 (15)
Sequestrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Serratia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 7 (7) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 2 (2)
Shoulder fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 4 (4)
Sinus node dysfunction (Cardiac disorders) | 7 (7) | 15 (15)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 10 (10) | 3 (3)
Skin oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (10)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleeve gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 10 (10) | 10 (12)
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 2 (2) | 0 (0)
Spermatic cord disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Spinal claudication (Nervous system disorders) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 8 (9) | 5 (5)
Spinal cord abscess (Infections and infestations) | 0 (0) | 1 (1)
Spinal cord infarction (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Squamoproliferative lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (8) | 3 (4)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (13) | 9 (10)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 3 (3)
Staphylococcal infection (Infections and infestations) | 3 (3) | 3 (3)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1)
Status migrainosus (Nervous system disorders) | 0 (0) | 1 (1)
Stent placement (Surgical and medical procedures) | 10 (10) | 12 (13)
Stent-graft endoleak (General disorders) | 2 (3) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Stoma obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Stress cardiomyopathy (Cardiac disorders) | 3 (3) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 6 (6) | 12 (12)
Subcapsular renal haematoma (Renal and urinary disorders) | 3 (3) | 0 (0)
Subclavian artery occlusion (Vascular disorders) | 1 (1) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 2 (2) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 16 (16) | 6 (6)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Subileus (Gastrointestinal disorders) | 0 (0) | 4 (4)
Subperiosteal abscess (Infections and infestations) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Sudden cardiac death (General disorders) | 8 (8) | 12 (12)
Sudden death (General disorders) | 5 (5) | 16 (16)
Sudden hearing loss (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 4 (5) | 4 (4)
Suicide attempt (Psychiatric disorders) | 1 (2) | 3 (3)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 18 (19) | 7 (7)
Suspected drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 65 (71) | 55 (63)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Systemic sclerosis pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 5 (5)
Takayasu's arteritis (Vascular disorders) | 1 (1) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 5 (6) | 6 (8)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 2 (2) | 0 (0)
Terminal ileitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Testicular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 4 (4)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 3 (3)
Thrombotic cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 3 (3)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis acute (Endocrine disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 9 (9)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Tissue infiltration (General disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 3 (5)
Toxic goitre (Endocrine disorders) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (2) | 4 (4)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tracheal compression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 2 (2)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 2 (2)
Transient aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 3 (3) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 39 (42) | 59 (63)
Transitional cell cancer of renal pelvis and ureter metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Transitional cell cancer of the renal pelvis and ureter localised (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 2 (2)
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic arthrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic heart injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic pancreatitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Treatment noncompliance (General disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 3 (3)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Troponin abnormal (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 3 (3)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 15 (15)
Type IIa hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Typical aura without headache (Nervous system disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 9 (9) | 4 (4)
Undifferentiated spondyloarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (13) | 14 (14)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urate nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 20 (21) | 10 (10)
Urethral meatus stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (2) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 4 (5) | 2 (2)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 5 (5)
Urinary retention (Renal and urinary disorders) | 11 (11) | 7 (7)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Urinary tract candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 32 (40) | 43 (46)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection pseudomonal (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 3 (3)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 14 (15) | 14 (15)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vagus nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Varicose ulceration (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 3 (3) | 2 (2)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 2 (2) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 2 (2)
Vascular device occlusion (General disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Vascular graft infection (Infections and infestations) | 1 (1) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 7 (11) | 8 (9)
Vascular graft restenosis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular occlusion (Vascular disorders) | 0 (0) | 2 (2)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 4 (5) | 4 (4)
Vascular stenosis (Vascular disorders) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 2 (2) | 8 (9)
Vascular stent stenosis (General disorders) | 22 (22) | 21 (25)
Vascular stent thrombosis (General disorders) | 1 (1) | 2 (2)
Venous thrombosis limb (Vascular disorders) | 2 (2) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 4 (4) | 4 (4)
Ventricular extrasystoles (Cardiac disorders) | 12 (12) | 9 (10)
Ventricular fibrillation (Cardiac disorders) | 7 (7) | 11 (12)
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 36 (36) | 38 (49)
Vertebral artery stenosis (Nervous system disorders) | 3 (3) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebrobasilar artery dissection (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 3 (3) | 2 (2)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 18 (18) | 7 (8)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 3 (3) | 7 (7)
Vestibular neuronitis (Infections and infestations) | 2 (2) | 2 (2)
Viral diarrhoea (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 4 (4)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 2 (2)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (18) | 12 (12)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 3 (3)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Wound infection pseudomonas (Infections and infestations) | 0 (0) | 2 (2)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 2 (2)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 2 (2) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (5)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 (1) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 1 (1)
Alcohol induced persisting dementia (Nervous system disorders) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Amaurosis (Eye disorders) | 1 (1) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 (0) | 1 (1)
Anti-thyroid antibody positive (Investigations) | 1 (1) | 0 (0)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bifascicular block (Cardiac disorders) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Body mass index increased (Investigations) | 0 (0) | 1 (1)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast reconstruction (Surgical and medical procedures) | 0 (0) | 1 (1)
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0)
Catatonia (Psychiatric disorders) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Central nervous system infection (Infections and infestations) | 1 (1) | 0 (0)
Cervix disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chordae tendinae rupture (Cardiac disorders) | 0 (0) | 1 (1)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Conjunctival neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dermatochalasis (Eye disorders) | 1 (2) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diffuse idiopathic skeletal hyperostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Eye haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 2 (2) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 1 (1) | 0 (0)
Gastric ulcer helicobacter (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Hashimoto's encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatobiliary procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Herpes simplex meningitis (Infections and infestations) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 2 (3)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 2 (4) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic mitral regurgitation (Cardiac disorders) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lenticular opacities (Eye disorders) | 1 (2) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphatic fistula (Vascular disorders) | 1 (2) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 1 (1) | 0 (0)
Motor neurone disease (Nervous system disorders) | 1 (1) | 0 (0)
Moyamoya disease (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1)
Myopia (Eye disorders) | 1 (1) | 0 (0)
Nasal abscess (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (2) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Normochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Orthostatic tremor (Nervous system disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Parotid abscess (Infections and infestations) | 1 (1) | 0 (0)
Pelvic floor dysfunction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Polyneuropathy alcoholic (Nervous system disorders) | 0 (0) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pseudoaneurysm (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Septic encephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Small intestine neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Spinal retrolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Superficial spreading melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Thalamic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ulcerative gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Vestibular ataxia (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Visual field defect (Eye disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Withdrawal catatonia (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide (N=8803) | Placebo (N=8801)
COVID-19 (Infections and infestations) | 1787 (1933) | 1785 (1935)
Constipation (Gastrointestinal disorders) | 715 (855) | 231 (256)
Decreased appetite (Metabolism and nutrition disorders) | 585 (655) | 112 (123)
Diarrhoea (Gastrointestinal disorders) | 933 (1417) | 353 (429)
Dyspepsia (Gastrointestinal disorders) | 468 (629) | 94 (102)
Nausea (Gastrointestinal disorders) | 1592 (2260) | 337 (414)
Vomiting (Gastrointestinal disorders) | 576 (752) | 87 (106)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03574597/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03574597/SAP_003.pdf